CLINICAL TRIAL: NCT02774629
Title: Efficacy of Local Lyophilized Food Extracts for Skin Prick Tests and Atopy Patch Test at Different Storage Times (0, 3 and 6 Months)
Brief Title: Efficacy of Local Food Extracts at Different Storage Times
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Other Study IDs: 619/2556(EC3)
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Food Allergy
Keywords: food allergy; skin prick test; atopy patch test
MeSH Terms: conditions — Food Hypersensitivity | interventions — Punctures; Patch Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: prick and patch test — The cases are pricked and patched with local food allergen extract at different storage times (0, 3 and 6 months after preparation)

SUMMARY:
Local lyophylized food extracts are available useful in skin prick test and atopy patch test to confirm food allergy. However, the investigators want to know the duration that the investigators can keep the extracts for the usage in this purpose.

DETAILED DESCRIPTION:
Food allergy incidence increases world wide. The diagnosis mostly depends on history. Skin prick test and atopic patch test are useful in finding the causative foods in some cases. The local food extracts have been shown to be at least as effective as commercial ones. From previous study the investigators keep the extract at 2-8 degree Celsius for 1-3 months for the usage. The investigators want to evaluate the duration that the extracts are still useful in diagnosis food allergy

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick test to one of the food (milk, egg, soy, wheat, seafood)

Exclusion Criteria:

* Chronic diseases such as heart disease, liver, renal and severe sepsis
* Severe allergic symptoms such as anaphylaxis
* Extensive skin rashes
* Pregnancy

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Food allergy cases aged 3-18 years old.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean wheal diameter of skin prick test | 2 years
  The skin prick tests are performed with local prepared food allergen at keeping time of 0, 3 and 6 months after the preparation.

SECONDARY OUTCOMES:
Result of atopy patch test | 2 years
  atopy patch tests are performed with local prepared food allergen at keeping time of 0, 3 and 6 months after the preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, Prof, Principal Investigator — Mahidol University
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No